CLINICAL TRIAL: NCT03657212
Title: Enhancing Memory Consolidation in Older Adults
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Changed University from UCR to UCI. The new lab was not adequately equipped to handle the sleep research and it was too far from the main lab. Funding was running out.
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Sara Mednick, Professor, University of California, Irvine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20184179
Record Dates: First submitted 2018-07-11; First posted 2018-09-04 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Aging
MeSH Terms: interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nap/5mg Zolpidem, then placebo (Experimental): The research involves oral administration of zolpidem (ZOL, 5mg) on week one and placebo on week two during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. The order of drug conditions will be randomized and counterbalanced. During the experimental phase, each drug condition will include one day in the sleep lab, two encoding test sessions, and one retrieval test session. Multiple subjects will be in the experimental phase concurrently, and multiple subjects will be tested on each day.
  Interventions: Drug: Zolpidem
- Nap/Placebo, then 5mg Zolpidem (Experimental): The research involves oral administration of placebo on week on and zolpidem (ZOL, 5mg) on week two during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. The order of drug conditions will be randomized and counterbalanced. During the experimental phase, each drug condition will include one day in the sleep lab, two encoding test sessions, and one retrieval test session. Multiple subjects will be in the experimental phase concurrently, and multiple subjects will be tested on each day.
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Drug: Zolpidem — The research involves oral administration of zolpidem (ZOL) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. One condition will be tested per week, with condition order counterbalanced. Each subject will have 2 visits (plus an adaptation nap), each separated by 5-7 days (although this may be extended based on participant availability) to ensure that the drug is completely eliminated from the body. The order of drug conditions will be randomized and counterbalanced.
  Other Names: Ambien; Edluar; Zolpimist

SUMMARY:
The purpose of this research study is to understand the neural mechanisms underlying long-term memory formation in older adults. Both sleep and memory decrease with age. The investigators are interested in discovering whether these two biological changes are related. This study is specifically focused on understanding what are the critical components of sleep that facilitate memory formation and are they impaired in older adults. The investigators will be using the hypnotic zolpidem, a sleep drug that has been shown to increase a specific aspect of sleep that have been shown to correlate with memory improvement in young adults. The Food and Drug Administration (FDA) have approved zolpidem for use in certain sleep disorders, specifically in the treatment of sleeplessness (i.e., insomnia). In the current study, the investigators will examine whether zolpidem (5mg), compared with placebo, increases memory-related sleep events in older adults and test the impact of these drug-related sleep changes on post-sleep memory recall.

This is a research study because the investigators are using pharmacological interventions to investigate our hypotheses about memory consolidation. The investigators are not studying the efficacy of zolpidem to treat conditions for which the FDA has already approved it.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* non-smoker
* between the ages of 60 to 75, without major medical problems
* have a regular sleep wake schedule, defined as obtaining 6-9 hours of sleep per night, with a habitual bedtime before 2am and a habitual wake time before 10am
* must have experience with Ambien to participate in the study.

Exclusion Criteria:

* have a sleeping disorder (reported or detected on questionnaires)
* have any personal or immediate family history of diagnosed mental disorders
* have any personal history of head injury with loss of consciousness greater than 2 minutes or seizures
* have a history of substance dependence
* currently use any medications that could affect sleep and/or thought processes
* have any cardiac, respiratory or other medical condition which may affect cerebral metabolism
* have dementia
* have non-correctable vision and hearing impairments, due to the nature of the stimulus and its presentation, will also be excluded.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara C Mednick, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- Sleep and Cognition Lab, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nap/5mg Zolpidem, Then Placebo; Nap/Placebo, Then 5mg Zolpidem: The research involves oral administration of zolpidem (ZOL, 5mg) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day.The order of drug conditions will be randomized and counterbalanced. During the experimental phase, each drug condition will include one day in the sleep lab, two encoding test sessions, and one retrieval test session. Multiple subjects will be in the experimental phase concurrently, and multiple subjects will be tested on each day.
  Zolpidem: The research involves oral administration of zolpidem (ZOL) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. One condition will be tested per week, with condition order counterbalanced. Each subject will have 2 visits (plus an adaptation nap), each separated by 5-7 days (although this may be extended based on participant availability) to ensure that the drug is completely eliminated from the body. The order of drug conditions will be randomized and counterbalanced.
Period: Overall Study
Arm/Group | Nap/5mg Zolpidem, Then Placebo | Nap/Placebo, Then 5mg Zolpidem
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Zolpidem Then Placebo; Placebo Then Zolpidem: The research involves oral administration of zolpidem (ZOL, 5mg) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day.The order of drug conditions will be randomized and counterbalanced. During the experimental phase, each drug condition will include one day in the sleep lab, two encoding test sessions, and one retrieval test session. Multiple subjects will be in the experimental phase concurrently, and multiple subjects will be tested on each day.
  Zolpidem: The research involves oral administration of zolpidem (ZOL) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. One condition will be tested per week, with condition order counterbalanced. Each subject will have 2 visits (plus an adaptation nap), each separated by 5-7 days (although this may be extended based on participant availability) to ensure that the drug is completely eliminated from the body. The order of drug conditions will be randomized and counterbalanced.
- Total: Total of all reporting groups
Arm/Group | Zolpidem Then Placebo | Placebo Then Zolpidem | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (4) | 60 (4) | 60 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Stanford Sleepiness Scale [Mean (Standard Deviation); unit: units on a scale] — Stanford Sleepiness scale is a scale from 1-10 with more sleepiness with higher numbers.
  units on a scale | 4.5 (1.5) | 5 (1.5) | 4.75 (1)
Epworth Sleepiness Scale [Mean (Standard Deviation); unit: units on a scale] — Epworth Measure is a measure of 1-15 with higher numbers indicating worse sleepiness.
  units on a scale | 11 (3) | 10 (3) | 10 (3)

OUTCOME MEASURES:

1. Primary Outcome: Memory Recall
Description: The investigators will assess change in performance on a memory task that will be tested before and after the drug intervention. Subjects will study word lists before the intervention and their recall will be tested after the intervention.
Time Frame: baseline to 12 hour recall test
Measure: Mean (Standard Deviation); unit: percent correct
Groups:
- Nap/5mg Zolpidem: This is data only for the zolpidem condition.
  The research involves oral administration of zolpidem (ZOL, 5mg) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. The order of drug conditions will be randomized and counterbalanced. During the experimental phase, each drug condition will include one day in the sleep lab, two encoding test sessions, and one retrieval test session. Multiple subjects will be in the experimental phase concurrently, and multiple subjects will be tested on each day.
  Zolpidem: The research involves oral administration of zolpidem (ZOL) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. One condition will be tested per week, with condition order counterbalanced. Each subject will have 2 visits (plus an adaptation nap), each separated by 5-7 days (although this may be extended based on participant availability) to ensure that the drug is completely eliminated from the body. The order of drug conditions will be randomized and counterbalanced.
- Nap/Placebo: This is data only for the placebo condition.
  The research involves oral administration of zolpidem (ZOL, 5mg) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. The order of drug conditions will be randomized and counterbalanced. During the experimental phase, each drug condition will include one day in the sleep lab, two encoding test sessions, and one retrieval test session. Multiple subjects will be in the experimental phase concurrently, and multiple subjects will be tested on each day.
  Zolpidem: The research involves oral administration of zolpidem (ZOL) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. One condition will be tested per week, with condition order counterbalanced. Each subject will have 2 visits (plus an adaptation nap), each separated by 5-7 days (although this may be extended based on participant availability) to ensure that the drug is completely eliminated from the body. The order of drug conditions will be randomized and counterbalanced.
Arm/Group | Nap/5mg Zolpidem | Nap/Placebo
Number analyzed (Participants) | 10 | 10
percent correct | 80 (3.5) | 81 (4.3)

2. Secondary Outcome: Electroencephalography (EEG) Activity During the Naps
Description: The investigators will measure electroencephalography (EEG) during the sleep, we are measuring spindle density, where higher density means more spindles. More spindles would be a sign of greater hippocampal memory consolidation.
Time Frame: second intervention occurs at least 7 days after the first intervention
Measure: Mean (Standard Deviation); unit: spindles per minutes
Groups:
- Nap/5mg Zolpidem: This is zolpidem only data.
  The research involves oral administration of zolpidem (ZOL, 5mg) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. The order of drug conditions will be randomized and counterbalanced. During the experimental phase, each drug condition will include one day in the sleep lab, two encoding test sessions, and one retrieval test session. Multiple subjects will be in the experimental phase concurrently, and multiple subjects will be tested on each day.
  Zolpidem: The research involves oral administration of zolpidem (ZOL) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. One condition will be tested per week, with condition order counterbalanced. Each subject will have 2 visits (plus an adaptation nap), each separated by 5-7 days (although this may be extended based on participant availability) to ensure that the drug is completely eliminated from the body. The order of drug conditions will be randomized and counterbalanced.
- Nap/Placebo: This is placebo only data.
  The research involves oral administration of zolpidem (ZOL, 5mg) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. The order of drug conditions will be randomized and counterbalanced. During the experimental phase, each drug condition will include one day in the sleep lab, two encoding test sessions, and one retrieval test session. Multiple subjects will be in the experimental phase concurrently, and multiple subjects will be tested on each day.
  Zolpidem: The research involves oral administration of zolpidem (ZOL) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. One condition will be tested per week, with condition order counterbalanced. Each subject will have 2 visits (plus an adaptation nap), each separated by 5-7 days (although this may be extended based on participant availability) to ensure that the drug is completely eliminated from the body. The order of drug conditions will be randomized and counterbalanced.
Arm/Group | Nap/5mg Zolpidem | Nap/Placebo
Number analyzed (Participants) | 10 | 10
spindles per minutes | 6 (3) | 5 (3.5)

ADVERSE EVENTS:
Time Frame: We collected adverse events over the three weeks that the subject was in the study.
Groups:
- Nap/5mg Zolpidem: This is data for zolpidem only.
  The research involves oral administration of zolpidem (ZOL, 5mg) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. The order of drug conditions will be randomized and counterbalanced. During the experimental phase, each drug condition will include one day in the sleep lab, two encoding test sessions, and one retrieval test session. Multiple subjects will be in the experimental phase concurrently, and multiple subjects will be tested on each day.
  Zolpidem: The research involves oral administration of zolpidem (ZOL) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. One condition will be tested per week, with condition order counterbalanced. Each subject will have 2 visits (plus an adaptation nap), each separated by 5-7 days (although this may be extended based on participant availability) to ensure that the drug is completely eliminated from the body. The order of drug conditions will be randomized and counterbalanced.
- Nap/Placebo: This is data for placebo only.
  The research involves oral administration of zolpidem (ZOL, 5mg) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. The order of drug conditions will be randomized and counterbalanced. During the experimental phase, each drug condition will include one day in the sleep lab, two encoding test sessions, and one retrieval test session. Multiple subjects will be in the experimental phase concurrently, and multiple subjects will be tested on each day.
  Zolpidem: The research involves oral administration of zolpidem (ZOL) or placebo during sleep with EEG recording. This study will employ a within-subject, crossover design, in which every subject experiences each of the following study conditions: Nap/5mg, Nap/placebo, plus an adaptation nap to be scheduled one week prior to the first experimental day. One condition will be tested per week, with condition order counterbalanced. Each subject will have 2 visits (plus an adaptation nap), each separated by 5-7 days (although this may be extended based on participant availability) to ensure that the drug is completely eliminated from the body. The order of drug conditions will be randomized and counterbalanced.
Arm/Group | Nap/5mg Zolpidem | Nap/Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Early termination was due to two issues. First, PI Mednick changed institutions from UC Riverside to UC Irvine. The transfer of the grant was significantly delayed. We ran out of the no-cost-extension funds. Second, even though the PI was assured that she could conduct pharmacology studies by her new institution, in actuality the research could not be conducted on the main campus, where the PI's lab was located. The PI found a Medical school location, but it was not feasible for sleep research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT03657212/Prot_001.pdf
  • Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT03657212/SAP_003.pdf
  • Informed Consent Form (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT03657212/ICF_000.pdf